CLINICAL TRIAL: NCT00658034
Title: Acupuncture for the Treatment of Chronic Post-Chemotherapy Fatigue: a Randomized Phase III Trial
Brief Title: Acupuncture for the Treatment of Chronic Post-Chemotherapy Fatigue
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alta Bates Summit Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08-IM-01
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Fatigue
Keywords: Cancer; Fatigue; Acupuncture
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Acupuncture
  Interventions: Procedure: Acupuncture
- 2 (Sham Comparator): Placebo Acupuncture
  Interventions: Procedure: Placebo Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Subjects will receive acupuncture weekly for six weeks. Subjects will complete a Brief Fatigue Inventory (BFI) questionnaire, a Functional Assessment of Cancer Treatment scale (FACT-G), and a Hospital Anxiety and Depression Scale(HADS) at week 7. The BFI and FACT-G will be repeated at week 8. At the end of the study, subjects will be asked to state whether they thought they were on true or placebo acupuncture and why.
  Arms: 1
Procedure: Placebo Acupuncture — Subjects will receive placebo acupuncture weekly for six weeks. During the placebo phase, placebo acupuncture needles will be applied a few mm away from the required points. The placebo acupuncture needle is a blunt tipped needle that moves up inside its handle. When it is pressed against the skin, the subject feels a slight prick and sees the handle of the needle moving towards the skin as if the needle has been inserted.
  Subjects will complete a BFI, a FACT-G, and a HADS at week 7. The BFI and FACT-G will be repeated at week 8. At the end of the study, subjects will be asked to state whether they thought they were on true or placebo acupuncture and why. Subjects in the placebo group will be given the option to receive true acupuncture.
  Arms: 2

SUMMARY:
This is a randomized, placebo controlled study in cancer patients reporting fatigue persisting for at least two months following completion of chemotherapy. Subjects will receive 6 weeks of either acupuncture or placebo treatment as a means of evaluating whether acupuncture reduces chronic fatigue after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-64 diagnosed with a malignancy (solid tumor or hematologic malignancy).
* Patients must have received chemotherapy.
* Patients must complain of fatigue following chemotherapy buy not prior to chemotherapy.
* At least 60 days must have elapsed between the last chemotherapy infusion and completion of the first baseline questionnaire.
* Mean baseline fatigue as measured by the Brief Fatigue Inventory must be four or above.

Exclusion Criteria:

* Anemia, defined as Hb<9 or active treatment for anemia. Iron supplementation is allowed as long as the dose has been stable for at least six weeks.
* Platelets less than 50,000/microliter or an Absolute Neutrophil Count less than 1,000/microliter.
* Baseline depression score on the Hospital Anxiety and Depression Scale of 11 or above, indicating clinical depression.
* Thyroid disorder, defined as either thyroid stimulating hormone or free T4 out of normal range, is excluded as it is a possible cause of fatigue unrelated to cancer therapy.
* Surgery under general anesthesia; immunotherapy; radiotherapy; or initiation of hormonal therapy within the three weeks prior to enrollment.
* Acupuncture in the previous six weeks.
* Change in use of any of the following drugs in the prior three weeks: opiates, antidepressants (other than selective serotonin reuptake inhibitors [SSRIs])/anxiolytics; OR change in use of SSRIs in the prior six weeks. "Change in use" is defined as initiation or cessation of treatment, or change in prescribed dose or regimen: changes in actual amounts of PRN medication taken are allowed.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether acupuncture reduces chronic fatigue after chemotherapy more effectively than placebo | six weeks

SECONDARY OUTCOMES:
To examine the long term effects of acupuncture treatment on fatigue | six months
To examine predictors of response to acupuncture treatment in terms of baseline symptoms, hemoglobin, age, sex, time since chemotherapy, and concurrent treatment | six months
To examine the effect of acupuncture on levels of physical activity and quality of life | six months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Matecki, MD, Principal Investigator — Alta Bates Summit Comprehensive Cancer Center
Locations (1):
- Alta Bates Summit Comprehensive Cancer Center, Berkeley, California, United States